CLINICAL TRIAL: NCT02225600
Title: The Effect of Oxytocin Administration on Interpersonal Cooperation in Borderline Personality Disorder Patients and Healthy Adults: A Pilot Behavioral Study
Brief Title: The Effect of Oxytocin Administration on Interpersonal Cooperation in Borderline Personality Disorder Patients and Healthy Adults
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Avoiding intranasal spray durng COVID
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Harold W Koenigsberg, MD, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: GCO 13-0744
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; BPD; Intranasal oxytocin
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients with BPD (Other): cross-over administration of 40 IU oxytocin, 24 IU oxytocin and placebo
  Interventions: Drug: 40 IU Intranasal Oxytocin; Drug: Placebo; Drug: 24 IU intranasal Oxytocin
- healthy patients (Active Comparator): Cross-over of 40 IU oxytocin, 24 IU oxytocin and placebo
  Interventions: Drug: 40 IU Intranasal Oxytocin; Drug: Placebo; Drug: 24 IU intranasal Oxytocin

INTERVENTIONS:
Drug: 40 IU Intranasal Oxytocin — 40 IU intranasal oxytocin
  Other Names: OT; Syntocin
Drug: Placebo — Intranasal Placebo
  Other Names: Intranasal Placebo
Drug: 24 IU intranasal Oxytocin
  Other Names: syntocin; OT

SUMMARY:
The study will examine behavioral patterns and underlying neural correlates which distinguish patients with borderline personality disorder (BPD) from healthy subjects as they participate in a two-person trust game and will determine whether administration of intranasal oxytocin (OT) will normalize trust game performance and concomitant neural processing in the BPD group.

DETAILED DESCRIPTION:
This is a pilot study to support submission of a larger-scale federally funded study. The study is designed to develop new strategies for treating the severe interpersonal dysfunction in borderline personality disorder (BPD) by modeling the interpersonal disturbance in BPD in the laboratory, identifying its neural correlates and determining whether the social neuropeptide, oxytocin, can ameliorate the interpersonal dysfunction. The study will examine behavioral patterns and underlying neural correlates which distinguish patients with borderline personality disorder (BPD) from healthy subjects as they participate in a two-person trust game and will determine whether administration of intranasal oxytocin (OT) will normalize trust game performance and concomitant neural processing in the BPD group.

The specific aims of the study are: 1) to determine whether BPD patients and healthy controls (HC) differ in their pattern of investing in a trustee when the trustee behaves benevolently or malevolently towards them or suddenly becomes malevolent after a period of benevolence (or vice-versa) in a multi-round economic exchange game ("The Trust Game"), and 2) to determine the effect upon behavior of the administration of 40 IU intranasal oxytocin relative to placebo in BPD subjects and HC's engaged in the Trust Game.

Subjects are being recruited and may participate in the Trust Game task, but intranasal administration of oxytocin has temporarily been held because of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* BPD subjects meets criteria for DSM-IV Borderline Personality Disorder.
* 18 to 55 years old
* Healthy controls are free of any lifetime DSM-IV Axis I or Axis II diagnosis. However, to avoid a group of HC's too highly groomed and unrepresentative of the general population subjects meeting criteria for a past Axis I diagnosis of adjustment, dysthymic, or depressive NOS disorders, specific phobias, and sleep disorders will not be excluded. Subjects will not be excluded for a non-IV substance abuse disorder more than 6 months prior to enrollment.
* All subjects will be free of psychotropic medications for 2 weeks (6 weeks for fluoxetine).
* Subjects may be enrolled in psychotherapy.

Exclusion Criteria:

* BPD subjects not meeting DSM-IV criteria for past or present bipolar I disorder, schizophrenia, schizoaffective disorder, substance dependence, head trauma, CNS neurological disease, seizure disorder or current major depression. Since depression is commonly associated with BPD, too stringent a depression exclusion criterion would yield a clinically atypical BPD sample. For this reason, BPD patients with Axis I depressive disorders other than major depression and those with a past history of major depression will not be excluded.
* Substance abuse disorder in the prior 6 months
* Significant medical illness
* Pregnancy
* Metallic foreign-bodies that contraindicate MRI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Trust Game Affect Ratings | up to 4 weeks
  Behavioral differences between groups based on Scale with 1= most negative to 5=most positive

CONTACTS AND LOCATIONS:
Overall Officials: Harold Koenigsberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States